CLINICAL TRIAL: NCT06045689
Title: A Phase 3b, Open-label Study Evaluating the Efficacy and Safety of Luspatercept (BMS-986346/ACE-536) Initiated at Maximum Approved Dose in LR-MDS With IPSS-R Very Low-, Low-, or Intermediate-risk Who Require RBC Transfusions (MAXILUS)
Brief Title: A Study to Assess Luspatercept in Lower-risk Myelodysplastic Syndrome Participants
Acronym: MAXILUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA056-1060
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Myelodysplastic Syndromes
Keywords: Luspatercept; Transfusion dependent; ACE-536; Anemia; Blood Transfusion; Red Blood Cell Transfusion; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: erythropoiesis-stimulating agents (ESA) naïve (Experimental)
  Interventions: Drug: Luspatercept
- Cohort 2: ESA relapsed or refractory (Experimental)
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Specified dose on specified days.
  Other Names: BMS-986346; ACE-536; REBLOZYL

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Luspatercept when administered at the maximum approved dose in low-risk Myelodysplastic Syndrome participants who require red blood cell transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Participant had documented diagnosis of MDS according to World Health Organization (WHO) classification that met Revised International Prognostic Scoring System (IPSS-R) classification of very low-, low-, or intermediate-risk disease.
* Participant has an Eastern Cooperative Oncology Group (ECOG) score of 0, 1, or 2.
* Participant must have red blood cell transfusions according to study criteria.

Exclusion Criteria:

* Participant has known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or gastrointestinal bleeding.
* Participant has had a prior allogeneic or autologous stem cell transplant.
* Participant has known history or diagnosis of AML.
* Participant has uncontrolled hypertension.

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve red blood cell transfusion independence (RBC-TI) for 8 weeks with a simultaneous mean hemoglobin (Hb) increase of ≥ 1 g/dL from Week 1 to Week 24 | Up to week 24

SECONDARY OUTCOMES:
Number of participants with a mean change in total RBC units transfused over a fixed 16-week period from Week 9 to Week 24 and from Week 33 to Week 48 | Up to week 48
Number of participants who have a time from first dose to first onset of RBC-TI ≥ 8-, 12-, and 16-weeks from Week 1 to Week 24, from Week 1 to Week 48, and from Week 1 through EOT | Up to 2 years
Number of participants who achieve RBC-TI over any consecutive 8-week period from Week 1 to Week 24, from Week 1 to Week 48, and from Week 1 to EOT | Up to 2 years
Number of participants with a maximum duration of RBC-TI for participants who achieve RBC TI ≥ 8- and 16-week period from Week 1 to Week 24 and from Week 1 to EOT | Up to 2 years
Number of participants who achieve RBC-TI over any consecutive 12-, 16-, and 24-week periods from Week 1 to Week 24, from Week 1 to Week 48 and from Week 1 through EOT | Up to 2 years
Number of participants with an increase from baseline in mean hemoglobin (Hb) values of ≥ 1.0 g/dL over any consecutive 8-week period in absence of RBC transfusions from Week 1 to Week 48 and from Week 1 through EOT | Up to 2 years
Number of participants with an increase from baseline in Hb values of ≥ 1.0 g/dL over any consecutive 16-week period in absence of RBC transfusions from Week 1 to Week 24, from Week 1 to Week 48, and from Week 1 through EOT | Up to 2 years
Number of participants with an increase from baseline in Hb values of ≥ 1.5 g/dL over any consecutive 8-, and 16-week periods in absence of RBC transfusions from Week 1 to Week 24, from Week 1 to Week 48, and from Week 1 through EOT | Up to 2 years
Number of participants who achieve Hematological Improvement Erythroid (mHI-E) per International Working Group-2018 (IWG-2018) over any consecutive 8-week period from Week 1 to Week 24, from Week 1 to Week 48, and Week 1 through EOT | Up to 2 years
Number of participants who achieve Hematological Improvement - Neutrophils (HI-N) per IWG-2018 over any consecutive 8-week period from Week 1 to Week 24, from Week 1 to Week 48, and Week 1 through EOT | Up to 2 years
Number of participants who achieve Hematological Improvement - Platelets (HI-P) per IWG-2018 over any consecutive 8-week period from Week 1 to Week 24, from Week 1 to Week 48, and Week 1 through EOT | Up to 2 years
Number of participants with change in serum ferritin (SF) over a 16-week period from Week 9 to Week 24 and from Week 33 to Week 48 | Up to week 48
Number of participants with change in mean daily dose of iron chelation therapy (ICT) over a 16-week period from Week 9 to Week 24 and from Week 33 to Week 48 | Up to week 48
Number of participants with adverse events (AEs) | Up to 2 years
Number of participants with acute myeloid leukemia (AML) progression | Up to 4 years
Time to AML progression | Up to 4 years
Time from treatment start date to death due to any cause | Up to 4 years
Number of participants with a change in subscale scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) from Week 1 to Week 48 and from baseline through EOT | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (52):
- United States (16):
  - Local Institution - 0051, Los Alamitos, California
  - Local Institution - 0033, New Haven, Connecticut
  - Local Institution - 0055, St. Petersburg, Florida
  - Local Institution - 0056, Wellington, Florida
  - Local Institution - 0020, Kansas City, Kansas
  - Local Institution - 0025, Paducah, Kentucky
  - Local Institution - 0011, Detroit, Michigan
  - Local Institution - 0059, St Louis, Missouri
  - Local Institution - 0058, Morristown, New Jersey
  - Local Institution - 0032, New York, New York
  - Local Institution - 0054, Eugene, Oregon
  - Local Institution - 0036, Pittsburgh, Pennsylvania
  - Local Institution - 0043, Amarillo, Texas
  - Local Institution - 0022, Huntsville, Texas
  - Local Institution - 0031, Wheeling, West Virginia
  - Local Institution - 0003, Milwaukee, Wisconsin
- Belgium (2):
  - Local Institution - 0016, Leuven, Vlaams Brabant
  - Local Institution - 0008, Roeselare, West-Vlaanderen
- Czechia (2):
  - Local Institution - 0023, Prague, Praha, Hlavní Mesto
  - Local Institution - 0004, Prague, Praha, Hlavní Mesto
- France (7):
  - Local Institution - 0041, Nice, Alpes-Maritimes
  - Local Institution - 0001, Poitiers, Vienne
  - Local Institution - 0026, Angers
  - Local Institution - 0007, Grenoble
  - Local Institution - 0046, Paris
  - Local Institution - 0053, Pierre-Bénite
  - Local Institution - 0044, Tour Cedex01
- Germany (3):
  - Local Institution - 0013, München, Bavaria
  - Local Institution - 0040, Hanover, Lower Saxony
  - Local Institution - 0009, Leipzig, Saxony
- Italy (8):
  - Local Institution - 0021, Reggio Calabria, Calabria
  - Local Institution - 0062, Napoli, Campania
  - Local Institution - 0050, Rome, Lazio
  - Local Institution - 0015, Pavia, Lombardy
  - Local Institution - 0029, Rozzano (MI), Milano
  - Local Institution - 0014, Novara, Piedmont
  - Local Institution - 0045, Turin, Piedmont
  - Local Institution - 0024, Florence, Tuscany
- Poland (4):
  - Local Institution - 0049, Lódz, Lódzkie
  - Local Institution - 0010, Warsaw, Masovian Voivodeship
  - Local Institution - 0034, Katowice
  - Local Institution - 0035, Wałbrzych
- Local Institution - 0047, San Juan, Puerto Rico
- Spain (9):
  - Local Institution - 0017, L'Hospitalet de Llobregat, Barcelona
  - Local Institution - 0005, Barcelona
  - Local Institution - 0052, Barcelona
  - Local Institution - 0039, Granada
  - Local Institution - 0038, Madrid
  - Local Institution - 0027, Ourense
  - Local Institution - 0028, Salamanca
  - Local Institution - 0018, Valencia
  - Local Institution - 0063, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06045689.html